CLINICAL TRIAL: NCT06528808
Title: The Effect of Simple Simulation-Based Breast Cancer Awareness Training on Women's Breast Cancer Knowledge and Fear Levels
Brief Title: Simple Simulation Based Breast Cancer Awareness Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBÜ-AYDINKARTAL-007
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer Awareness Training
Keywords: Simulation Based; Breast Cancer Awareness

STUDY DESIGN:
Intervention Model Description: Quasi-experimental randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (n:40) (Experimental): Women in the intervention group will undergo a simulator breast cancer awareness application in simple reality.
  Interventions: Other: Simple reality simulator application
- Control group (n:40) (No Intervention): Control group women will receive 2 hours of theoretical training.

INTERVENTIONS:
Other: Simple reality simulator application — Women in the intervention group will be given an application aimed at breast cancer awareness with a simple valid simulator.
  Arms: İntervention group (n:40)

SUMMARY:
It was planned to determine the effect of simple simulation-based breast cancer awareness training on women's breast cancer knowledge and fear levels. The research population will consist of female service personnel working in institutions within the University of Health Sciences (SBÜ) (N: 670). In order to determine the sample size in this research, which was planned as a quasi-experimental with a pre- and post-test design and a control group; The data showed a normal distribution, the standard deviation of the population was estimated to be 1, and the effect size (difference) was estimated to be 0.8. It was calculated that if two independent n₁=40, n₂=40 samples were taken for the analysis to be carried out, at a 5% significance level, the maximum power value of the research would be 0.942182. Both groups will be given theoretical training about breast cancer awareness, and women in the intervention group will practice breast cancer awareness with a simple valid simulator. All groups will be informed before the applications. The training content will be supported by distributing a 5-page training booklet created from breast health and cancer awareness content to the participants. "Comprehensive Breast Cancer Knowledge Test", "Breast Cancer Fear Scale" and "Breast Cancer Awareness Scale" will be applied as a pre-test after the information.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research.
* To work as female service personnel in institutions within the University of Health Sciences.

Exclusion Criteria:

- Not participating in all applications of simulation teaching.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 10 minutes
  In this form, created by the researchers based on the literature, participants' age, obstetric history (number of pregnancies, number of births, breastfeeding status, etc.), self-breast examination status, etc. questions are included.
Comprehensive Breast Cancer Knowledge Test | 10 minutes
  The scale, developed by Stager in 1993, consists of 20 knowledge questions. The Turkish adaptation of the scale was carried out by Başak and Tosun in 2015. The scale is answered in a true-false manner, and there are 8 correct and 12 incorrect answers among the questions. After the test application is carried out; According to the answer key of the scale, "correct" answers are given 1; "Incorrect" and blank answers were given 0 points. GKMKBT includes two dimensions: general knowledge and treatability. Questions from 1 to 12; general knowledge about breast cancer; Questions 13 to 20 contain information about the treatability of breast cancer. The reliability of the scale was found to be 0.71.
Breast Cancer Fear Scale | 10 minutes
  It was developed by Champion in 2004 to examine women's breast cancer fears by determining their emotional responses to breast cancer and screening. The Turkish validity and reliability study of the scale was conducted by Seçginli in 2012. The scale contains eight items and is scored on a 5-point Likert type. According to this scoring, the lowest possible score is 8 and the highest score is 40. A higher score from the scale indicates a higher level of breast cancer fear. On scale; Scoring between 8 and 15 indicates a low level of fear of breast cancer, scoring between 16 and 23 indicates a moderate level of fear of breast cancer, and scoring between 24 and 40 indicates a high level of fear of breast cancer. Cronbach's Alpha value of the scale was found to be 0.90.
Breast Cancer Awareness Scale | 10 minutes
  The scale was developed in 2010 by the UK cancer research center, "King's College London" and "University College London" to determine breast cancer awareness. In our country, the Turkish validity and reliability study of the scale was conducted by Baş and Ursavaş (2022). The scale consists of a total of 13 items to determine breast cancer awareness, including symptoms (11 items), frequency of breast examination (1 item) and breast cancer age (1 item). The scale has no cut-off point. Answering 5 of the symptoms correctly is coded as 1 point, a 70-year-old woman is coded as 1 point, and breast examination once a month is coded as 1. Incorrect answers are worth 0 points. Scoring is between 0-3. Cronbach's alpha value of the scale was found to be 0.89. As the score obtained from the scale increases, breast cancer awareness increases.

SECONDARY OUTCOMES:
Comprehensive Breast Cancer Knowledge Test | 10 minutes
  The scale, developed by Stager in 1993, consists of 20 knowledge questions. The Turkish adaptation of the scale was carried out by Başak and Tosun in 2015. The scale is answered in a true-false manner, and there are 8 correct and 12 incorrect answers among the questions. After the test application is carried out; According to the answer key of the scale, "correct" answers are given 1; "Incorrect" and blank answers were given 0 points. GKMKBT includes two dimensions: general knowledge and treatability. Questions from 1 to 12; general knowledge about breast cancer; Questions 13 to 20 contain information about the treatability of breast cancer. The reliability of the scale was found to be 0.71.
Breast Cancer Fear Scale | 10 minutes
  It was developed by Champion in 2004 to examine women's breast cancer fears by determining their emotional responses to breast cancer and screening. The Turkish validity and reliability study of the scale was conducted by Seçginli in 2012. The scale contains eight items and is scored on a 5-point Likert type. According to this scoring, the lowest possible score is 8 and the highest score is 40. A higher score from the scale indicates a higher level of breast cancer fear. On scale; Scoring between 8 and 15 indicates a low level of fear of breast cancer, scoring between 16 and 23 indicates a moderate level of fear of breast cancer, and scoring between 24 and 40 indicates a high level of fear of breast cancer. Cronbach's Alpha value of the scale was found to be 0.90.
Breast Cancer Awareness Scale | 10 minutes
  The scale was developed in 2010 by the UK cancer research center, "King's College London" and "University College London" to determine breast cancer awareness. In our country, the Turkish validity and reliability study of the scale was conducted by Baş and Ursavaş (2022). The scale consists of a total of 13 items to determine breast cancer awareness, including symptoms (11 items), frequency of breast examination (1 item) and breast cancer age (1 item). The scale has no cut-off point. Answering 5 of the symptoms correctly is coded as 1 point, a 70-year-old woman is coded as 1 point, and breast examination once a month is coded as 1. Incorrect answers are worth 0 points. Scoring is between 0-3. Cronbach's alpha value of the scale was found to be 0.89. As the score obtained from the scale increases, breast cancer awareness increases.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No